CLINICAL TRIAL: NCT06691867
Title: Integrative Strong Body and Mind Training for Pediatric Sickle Cell Pain (I-STRONG for SCD): Multi-site, Randomized Clinical Trial
Brief Title: Integrative Training Program for Pediatric Sickle Cell Pain
Acronym: I-STRONG SCD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Soumitri Sil, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY00008060; R33AT012421 (NIH); 2024P007498 (Other: Emory IRB)
Record Dates: First submitted 2024-11-13; First posted 2024-11-18 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Pain; Lifestyle considerations; Pediatrics; Behavioral intervention; Mind-body intervention
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- I-STRONG - Early Start (Experimental): Youth and caregivers will receive the I-STRONG for SCD intervention in addition to standard care.
  Interventions: Behavioral: I-STRONG
- Enhanced Usual Care (EUC) (Other): Participants randomized to EUC will continue with standard care and optimal management of their SCD and chronic pain for approximately 8 months. After completing the 6-month follow-up assessment, participants will have the opportunity to start the I-STRONG SCD intervention.
  Interventions: Other: Enhanced Usual Care (EUC)

INTERVENTIONS:
Behavioral: I-STRONG — I-STRONG is an evidence-based protocol from the FIT Teens program. This intervention combines mind-body and cognitive-behavioral approaches with neuromuscular movement training informed by pediatric sports medicine and injury prevention research. It aims to teach mind-body skills applicable during movement training to enhance psychological coping and reduce fear of pain and activity avoidance.
  I-STRONG consists of 16 group-based telehealth sessions held twice weekly over 8 weeks. Each group can accommodate up to 6 patients with SCD. Adolescents are expected to attend all sessions, while parents will attend 6 of the 16. Parents will receive education about I-STRONG, guidance on supporting their teen's behavior change, and opportunities for networking with other parents of youth with SCD. Sessions will include brief daily homework (e.g., using phone apps to practice skills) to facilitate proficiency. Participants will self-report their practice of assigned skills.
  Other Names: Intervention Group
  Arms: I-STRONG - Early Start
Other: Enhanced Usual Care (EUC) — The EUC arm is designed to account for potential effects on time and standard medical care outcomes. Patients randomized to EUC will continue with standard care and optimal management of their SCD and chronic pain for approximately 8 months (i.e., time from enrollment through 6-month post-treatment assessment) before starting the intervention program to coincide with the study duration of the ES arm. After completing the 6-month follow-up assessment, patients will have the opportunity to start the I-STRONG for SCD intervention.
  Other Names: Control Group
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
This research aims to answer the question: does a group training program specifically for teens with chronic sickle cell disease (SCD) pain that teaches skills to strengthen the mind and body help improve everyday functioning and reduce pain symptoms?

The program will be tailored to address challenges related to frequent or chronic sickle cell pain and may improve participants' physical and emotional health.

The program, called I-STRONG for SCD (Integrative Strong Body and Mind Training for Sickle Cell Disease), may help improve everyday functioning and pain symptoms in teens with chronic pain related to SCD. The research team aims to determine how participants (teens and parents) respond to this program.

DETAILED DESCRIPTION:
I-STRONG for SCD integrates evidence-based mind-body, cognitive-behavioral, and neuromuscular movement training. It will be tested using an individually randomized group treatment (IRGT) design, comparing early start to the enhanced usual care. The primary objective is to determine whether I-STRONG for SCD combined with standard care is more effective than standard care alone in improving pain intensity from baseline to the 3-month follow-up in adolescents with SCD.

Adolescent participants with sickle cell disease and their caregivers will be recruited for this study. Participants of all genders, races, and ethnicities are eligible, with a majority expected to be Black or African American females, consistent with previous studies of individuals with SCD and chronic pain. The study will last approximately 36 months, with participant involvement lasting 9 months.

I-STRONG for SCD has been adapted from the Fibromyalgia Integrative Training for Teens (FIT Teens) program based on feedback from patients and caregivers, focusing on chronic SCD pain. In addition to usual care, participants will receive the I-STRONG intervention, which consists of 16 group-based telehealth sessions (90 minutes each), held twice weekly for 8 weeks. All patients can participate in I-STRONG, with randomization determining whether they begin with Early Start (after completing the baseline assessment) or Enhanced Usual Care (approximately 8 months after the baseline assessment).

Support from and inclusion in the National Institutes of Health (NIH) Helping to End Addiction Long-term Initiative (HEAL), or NIH HEAL Initiative, is provided for this study. For more information about the initiative visit the HEAL Initiative (https://heal.nih.gov/).

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form for adolescents 18 years old and caregivers' participation
* For children <18, informed assent and parental informed consent to participate in the study
* Willingness to comply with all study procedures and lifestyle considerations and availability for the duration of the study
* Males and females; Ages 12-18 years for adolescents; no age limitations for caregivers
* Documented diagnosis of sickle cell disease (any genotype) for adolescents
* Adolescent scores at least 3 on the Pediatric Pain Screening Tool
* Adolescent reports typical pain intensity in the past week at least 4 on a 0-10 cm Visual Analog Scale
* Adolescent on stable disease-modifying treatments, if applicable (e.g., hydroxyurea, glutamine, voxelotor, crizanlizumab) as defined by not newly initiated or significantly increased dosages (mg/kg) in the past 3 months
* Speak and read English

Exclusion Criteria:

* An adolescent has comorbid medical conditions typically associated with pain but unrelated to SCD (e.g., rheumatologic disorders or inflammatory bowel disease)
* Adolescent has undergone genetic or hematopoietic stem cell therapy
* Presence of a condition(s) or diagnosis, either physical or psychological, or physical exam finding that precludes participation
* Adolescents receiving active treatment (e.g., weekly appointments with a provider) for nonpharmacological therapies (e.g., structured behavioral pain management, physical therapy, or acupuncture program) that overlap with the active phase of the study intervention

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 155 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) Pain severity | Baseline, immediately post-intervention, 3 months and 6 months post-intervention
  Pain intensity is rated with the pain severity item of the Brief Pain Inventory (BPI). The single item is scored on a scale from 0 to 10 where no pain = 0 and severe pain = 10.
  This outcome applies to teens only.

SECONDARY OUTCOMES:
Change in Brief Pain Inventory (BPI) Pain Interference Score | Baseline, immediately post-intervention, 3 months and 6 months post-intervention
  Functional interference due to pain rated with the impact of pain on daily functions item of the Brief Pain Inventory (BPI). The single item is scored on a scale from 0 to 10 where no pain = 0 and severe pain = 10.
  This outcome applies to teens only.
Patient Health Questionnaire (PHQ-8) Score | Baseline, immediately post-intervention, 3 months and 6 months post-intervention
  Depressive symptoms in past two weeks among teen study participants and parents is assessed with the Patient Health Questionnaire (PHQ-8). The PHQ-8 has 8 items that are responded to on a 4-point scale where " not at all" = 0 and "nearly every day" = 3. Total scores range from 0 to 24 where higher scores indicate increased symptoms of depression.
  The outcome applies to teens and parents.
General Anxiety Disorder (GAD-2) | Baseline, immediately post-intervention, 3 months and 6 months post-intervention
  General worry in the past two weeks among teen study participants and parents will be assessed using the GAD-2 instrument. The GAD-2 has 2 items that are responded to on a 4-point scale where " not at all" = 0 and "nearly every day" = 3. Total scores range from 0 to 6 where higher scores indicate increased experiences of worry.
  The outcome applies to teens and parents.
Pain Catastrophizing Scale | Baseline, immediately post-intervention, 3 months and 6 months post-intervention
  Exaggerated worried thoughts of pain will be assessed among teen study participants and parents. The Pain Catastrophizing Scale, Child and Parent Report, is a 13-item well-validated self-report and parent-report measure of worried thoughts about pain. Items are answered on a 5-point scale where 0 = not true at all and 4 = very true. Total scores range from 0 to 52 and higher scores indicate increased catastrophic thinking.
  The outcome applies to teens and parents.
Pediatric Quality of Life Inventory (PedsQL) Score | Baseline, immediately post-intervention, 3 months and 6 months post-intervention
  Health-related quality of life and impact on child and family in the past month is assessed among teen study participants and parents with the Pediatric Quality of Life Inventory (PedsQL). The 23-item PedsQL was developed as part of the NIH Roadmap Initiative to create universal measures for patient-reported outcomes and contains questions in the domains of social peer, depression, anxiety, mobility, and function. Responses are given on a 5-point scale where 0 = never and 4 = almost always. Items are reverse scored and linearly transformed to a scale of 0 to 100, where higher total mean scores indicate a better quality of life.
  The outcome applies to teens only.
Adolescent Sleep-Wake Scale (ASWS) Score Short Form | Baseline, immediately post-intervention, 3 months and 6 months post-intervention
  The Adolescent Sleep Wake Scale (ASWS) Short Form is a 14-item patient report describing the occurrence and frequency of various behavioral sleep characteristics over the past month. Responses are given on a 6-point Likert scale where 1 = always and 6 = never. Total scores range from 14 to 84 and higher scores indicate better sleep quality.
  This outcome applies to teens only.
National Institute on Drug Abuse (NIDA)-Modified ASSIST (NM ASSIST) Tool Level 2 score | Baseline, 3 months post-intervention
  Substance use among teen study participants during the past 3 months is assessed with the NIDA-Modified Assist Tool Level 2 for children aged 11-17. The instrument asks respondents how often they have used 15 different substances. Responses are given on a 4-point scale where "not at all" = 0 and "nearly every day" = 4. The tool is scored as the number of items with a score greater than 0 and multiple items with scores above 0 indicate increased substance use.
  This outcome applies to teens only.
Opioid Use | Baseline, immediately post-intervention, 3 months and 6 months post-intervention
  Daily use of opioid pain medication will be determined based on participant completion of daily diaries for 1-week at each assessment visit. Participants will record opioid use daily (yes/no).
Opioid morphine milligram equivalent Use | Baseline and 3 months post-intervention
  An electronic medical chart review will determine opioid morphine milligram equivalent (MME) calculation in the past month, with higher scores indicating higher MME per day.
Patient Global Impression of Change (PGIC) Score | Baseline, 3 months and 6 months post-intervention
  The overall self-reported rating of the treatment's efficacy will be assessed with the Patient's Global Impression of Change (PGIC) instrument. The PGIC asks respondents to rate their overall improvement compared to the baseline. Responses are indicated on a scale of 1 to 7, where 1 = very much improved and 7 = very much worse.
  This outcome applies to teens only.
Treatment Evaluation Inventory-Short Form (TEI-SF) Score | Immediately post-intervention
  Teens and parents will complete the Treatment Evaluation Inventory-Short Form at the end of treatment. This form includes 9 items adapted to be specific to pediatric pain. Items are rated on a 5-point Likert scale ranging from 1 to 5. Total scores range from 9 to 45. Higher scores indicate increased acceptability with the study treatment.
  This outcome applies to teens and parents
Tampa Scale of Kinesiophobia (TSK) Score | Baseline, immediately post-intervention, 3 months and 6 months post-intervention
  Fear of movement related to fear of pain is assessed with the Tampa Scale of Kinesiophobia (TSK) instrument. The TSK is a 17-item questionnaire where responses are given on a 4-point Likert scale. Responses of "strongly agree" are coded as 1 and responses of "strongly agree" are coded as 4. Total scores range from 17 to 68 where higher scores indicate greater kinesiophobia.
  This outcome applies to teens only.
PROMIS Pediatric Fatigue Short Form | Baseline, immediately post-intervention, 3 months and 6 months post-intervention
  Perceptions of a child's tiredness and energy will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Fatigue Short Form. It consists of 10 items scored on a Likert-type scale ranging from 1 (never) to 5 (almost always). The total possible range is 10-50, with higher scores representing greater fatigue or lower energy, while lower scores indicate better energy levels or less fatigue.
  The outcome applies to teens and parent-proxy.
Chronic Pain Acceptance Questionnaire (CPAQ) | Baseline, immediately post-intervention, 3 months and 6 months post-intervention
  The 20-item CPAQ-revised has been designed to measure acceptance of pain. The acceptance of chronic pain is thought to reduce unsuccessful attempts to avoid or control pain and thus focus on engaging in valued activities and pursuing meaningful goals. The items on the CPAQ are rated on a 7-point scale from 0 (never true) to 6 (always true). To score the CPAQ, the Activity engagement and Pain willingness items are added to obtain a score for each factor. All the scores for each factor are summed to get the total score. Higher scores indicate higher levels of acceptance.
  The outcome applies to teens only.
Coping Self-Efficacy | Baseline, immediately post-intervention, 3 months and 6 months post-intervention
  The Child Self-Efficacy Scale (CSES) is a self-report tool that examines self-efficacy despite pain to assess normal functioning and behavior. The CSES is a 7-item form asking how sure a child can perform certain activities while in pain. An 11-point scale with anchor points being 0 (cannot do at all), 5 (moderately certain can do), and 10 (certain can do). A higher score suggests that a person is more confident in their ability to cope and function with pain.
  The outcome applies to teens and parent-proxy.
Therapeutic Factor Inventory - 8 (TFI-8) | Immediately post-intervention
  TFI-8 is a brief, reliable, and valid measure used for continuous process measurement and feedback to improve the functioning of therapy groups. The TFI-8 is given to participants after group therapy sessions to assess group cohesion. It typically consists of 8 items that respondents rate based on their experiences. Participants usually respond using a Likert scale (e.g., 1 to 5), where 1 may indicate "strongly disagree" and 5 indicates "strongly agree." The total score is calculated by summing the responses for all items. Higher total scores generally indicate a greater presence of therapeutic factors perceived by the participants.
  The outcome applies to teens only.

CONTACTS AND LOCATIONS:
Overall Officials: Soumitri Sil, PhD, ABPP, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Arthur M. Blank Hospital | Children's Healthcare of Atlanta, Atlanta, Georgia
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data will be available for sharing including study-level metadata and NIH Helping to End Addiction Long-term (HEAL) Common Data Elements.
Supporting Information: Study Protocol
Time Frame: Data will be available for sharing beginning 9 months and ending 36 months following article publication.
Access Criteria: Data for sharing will be available in an NIH HEAL-approved data repository for public use.